CLINICAL TRIAL: NCT02370004
Title: FASTA: Flexibility and Strength Training in Asthma
Brief Title: Flexibility and Strength Training in Asthma
Acronym: FASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director, Asthma Research Center, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014p000994
Record Dates: First submitted 2014-09-02; First posted 2015-02-24 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Asthma
Keywords: Asthma; RFST; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistive Flexibility and Strength Training (Experimental): Each subject will undergo Resistive Flexibility and Strength Training (RFST) with a trained practitioner.
  Interventions: Procedure: Resistive Flexibility and Strength Training

INTERVENTIONS:
Procedure: Resistive Flexibility and Strength Training — RFST is a physical therapy technique where a certified practitioner extends or flexes a joint with the subject actively resists the motion applied by the practitioner.
  During the RFST treatment a subject will lie on a massage table while the practitioner holds the subject's arm or leg and flexes or extends the limb, instructing the patient to resist the flexion or extension produced by the practitioner. The process is repeated a number of times for each muscle while varying joint positions.

SUMMARY:
The aim of the study is proof of concept and to establish the feasibility of performing a study of resistive flexibility and strength training (RFST) in patients with asthma, with the future goal of designing a larger randomized trial to test the hypothesis that RFST leads to greater improvement in asthma symptoms, pulmonary function tests, range of motion and connective tissue mobility compared with a control conventional physical therapy intervention.

DETAILED DESCRIPTION:
The treatment of symptomatic asthma currently focuses on the use of medications - inhaled or systemic - that have the principal goals of relieving airway pathology, namely airway narrowing, inflammation, mucus metaplasia and hyper-reactivity. There are no therapies directed at the chest wall or its connective tissue structural units, including connective tissue matrix, bone health and chest wall musculature. Resistive flexibility and strength training (RFST) is a new physical therapy technique that has successfully addressed abnormalities in the upper and lower extremities and back. In this application, we propose to use internal funding for a pilot project to explore the potential holistic benefits of RFST directed to the chest wall in symptomatic asthmatics as well as the potential mechanical basis of its therapeutic benefits if observed.

In RFST, the practitioner extends or flexes a joint, while the patient actively resists the motion applied by the practitioner. In other words, the patient performs an eccentric contraction of extensor muscles if the joint is flexed, or of flexor muscles if the joint is extended. The technique is based on the following theoretical principles:

* Opposing muscle pairs (i.e. ipsilateral flexor/extensor) can become dysfunctional when connective tissue within one of the muscles (either the flexor or the extensor) becomes chronically shortened-thought to be due to long-standing exaggerated centrally driven tonic muscle activity either following an injury or due to posture habit. When this happens, connective tissue within the opposing muscle will become chronically lengthened due to shortening of the paired muscle.
* The connective tissue can become inelastic and restrictive resulting in the muscles being held in a chronically short or lengthened position. These positions can change.
* In the trunk, imbalances can occur between flexor/extensor groups (e.g. psoas/multifidus) and also between right/left muscle pairs, creating postural asymmetries. For example, shortening of the psoas muscle on one side will lead to lengthening of the psoas on the contralateral side.
* Shortening of limb girdle muscles (e.g. pectoralis, gluteus) can create complex imbalance patterns both across local flexor/extensor pairs, across sides, and diagonally across the trunk (e.g. shortening of pectoralis major on one side causing lengthening of extensor muscles in contralateral hip).
* The end result of these imbalances is that the shortened muscles restrict the range of movement, and the lengthened muscles cannot function optimally in a lengthened position.

It is thought that resistance stretching 1) allows the shortened muscles to lengthen and the lengthened muscles to shorten by remodeling intramuscular and perimuscular connective tissue, 2) allows lengthened muscles to contract at a more favorable length and 3) allows for an increase in flexion, extension, and flexibility through joint ranges of motion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age ≥ 18 yrs
* Physician-diagnosed asthma
* Currently taking asthma medications
* Asthma Control Questionnaire (ACQ) score >1.25

Exclusion Criteria:

* Smoking history of ≥10 pack years
* Pregnancy or lactation or subjects planning to get pregnant during the course of the trial
* Major medical problems prohibiting study participation, i.e. presence of chronic or active lung disease other than asthma or history of unstable significant medical illness other than asthma or concurrent medical problems that would place the participant at increased risk as determined by the study physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Resistive Flexibility and Strength Training: Each subject will undergo Resistive Flexibility and Strength Training (RFST) with a trained practitioner.
  Resistive Flexibility and Strength Training: RFST is a physical therapy technique where a certified practitioner extends or flexes a joint with the subject actively resists the motion applied by the practitioner.
  During the RFST treatment a subject will lie on a massage table while the practitioner holds the subject's arm or leg and flexes or extends the limb, instructing the patient to resist the flexion or extension produced by the practitioner. The process is repeated a number of times for each muscle while varying joint positions.
Period: Overall Study
Arm/Group | Resistive Flexibility and Strength Training
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Resistive Flexibility and Strength Training
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 22.8 [19 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume at One Second - FEV1 % Predicted
Description: Forced expiratory volume - an assessment of pulmonary function
Time Frame: Change from baseline to end of study - 5 weeks
Measure: Mean (95% Confidence Interval); unit: % predicted
Arm/Group | Resistive Flexibility and Strength Training
Number analyzed (Participants) | 10
% predicted
  Pre Intervention | 91.4 [81.6 to 97.3]
  Post Intervention | 93.4 [83.6 to 99.3]
Statistical Analysis 1: Comparison: Resistive Flexibility and Strength Training; Paired T-tests were used to evaluate changes in spirometry results; Test type: Other; p = .10, t-test, 2 sided

2. Secondary Outcome: Asthma Control Test (ACT)
Description: Asthma Control Test is a questionnaire that assesses asthma control by asking about asthma symptoms during the last month.
  The minimum score is 5 and the maximum is 25. Any score <20 represents asthma that is not well controlled, the lower the number the worse the control.
Time Frame: Change from baseline to end of study - 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Asthma Control Test: Asthma Control Test which is a measure of asthma control and symptoms over the last four weeks
Arm/Group | Asthma Control Test
Number analyzed (Participants) | 10
units on a scale
  Pre Intervention | 19.2 (3.3)
  Post Intervention | 21.2 (1.5)

3. Secondary Outcome: Range of Motion Measurement- Circumference
Description: Range of motion measurements will help to assess the effectiveness of resistive flexibility and strength training. Circumference was measured using centimeters
Time Frame: Change from baseline to end of study - 5 weeks
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Range of Motion- Pre Intervention- Circumference: Range of Motion and mobility- pre intervention
- Range of Motion- Post Intervention- Circumference: Range of Motion - Post intervention
Arm/Group | Range of Motion- Pre Intervention- Circumference | Range of Motion- Post Intervention- Circumference
Number analyzed (Participants) | 10 | 10
cm
  Chest Circumference at Armpits, inhalation | 93.1 (8.3) | 95.4 (8.8)
  Chest Circumference at Armpits, exhalation | 88.9 (8.4) | 90.4 (9.3)
  Chest Circumference at Xiphoid, inhalation | 78.7 (7.2) | 82.4 (8.7)
  Chest Circumference at Xiphoid, exhalation | 75.3 (9.2) | 77.6 (9.7)

4. Secondary Outcome: Range of Motion Measurements- Degree of Motion
Description: Range of motion measurements will help to assess the effectiveness of resistive flexibility and strength training. Range of motion was measured using degrees
Time Frame: Change from baseline to end of study- 5 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Range of Motion- Pre Intervention- Degree: Range of Motion and mobility- pre intervention
- Range of Motion- Post Intervention- Degree: Range of Motion - Post intervention
Arm/Group | Range of Motion- Pre Intervention- Degree | Range of Motion- Post Intervention- Degree
Number analyzed (Participants) | 10 | 10
Degrees
  FMS Shoulder Mobility Left | 8.5 (7.0) | 8.5 (8.8)
  FMS Shoulder Mobility Right | 9.6 (9.4) | 8.1 (7.8)
  Posterior Arm Extension Left | 37.6 (7.5) | 38.7 (9.7)
  Posterior Arm Extension Right | 34.9 (8.8) | 39.7 (10.0)
  Arm Raise Left | 151.0 (22.7) | 165.4 (18.3)
  Arm Raise Right | 154.1 (21.1) | 165.6 (20.9)

ADVERSE EVENTS:
Arm/Group | Resistive Flexibility and Strength Training
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No